CLINICAL TRIAL: NCT04661007
Title: A Phase 1b/2 Study of Tafasitamab, Tafasitamab Plus Lenalidomide, Tafasitamab Plus Parsaclisib, and Tafasitamab Plus Lenalidomide in Combination With R-CHOP in Japanese Participants With Non-Hodgkin Lymphoma
Brief Title: To Assess the Safety and Tolerability of Tafasitamab Alone or in Combination With Other Drugs in Japanese Participants With Non-Hodgkins Lymphoma (NHL)
Acronym: J-MIND
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Incyte Biosciences Japan GK (Industry)
Responsible Party: Sponsor
Organization: Incyte Corporation (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCMOR 0208-102
Record Dates: First submitted 2020-12-01; First posted 2020-12-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Non Hodgkins Lymphoma; Diffuse Large B-cell Lymphoma
Keywords: INCMOR00208; tafasitamab
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse | interventions — tafasitamab; Lenalidomide; parsaclisib; R-CHOP protocol

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Part 1 : tafasitimab monotherapy (Experimental): Dose-finding to evaluate the safety and tolerability and to determine the RP2Ds of single-agent tafasitamab in Japanese participants with NHL. Part 1 consists of 1 group (Group 1) to evaluate weight-based doses of tafasitamab.
  Interventions: Drug: tafasitamab
- Part 2 : tafasitamab combination therapy (Experimental): tafasitamab will be combined with lenalidomide (Group 3) or parsaclisib (Group 4a) in R/R DLBCL participants or lenalidomide plus R-CHOP (Group 5) in previously untreated DLBCL participants. Modified tafasitamab dosing when combined with lenalidomide (Group 2) in participants with R/R DLBCL will be evaluated to determine the recommended clinical dose. The dose of tafasitamab will be based on the weight-based RP2D that is deemed safe and tolerable in Part 1.
  Interventions: Drug: tafasitamab; Drug: lenalidomide; Drug: parsaclisib; Drug: R-CHOP
- Part 3 : Dose Expansion of tafasitamab +parsaclisib (Experimental): tafasitamab in combination with parsaclisib will be further evaluated in Group 4b at RP2D determined in Part 2
  Interventions: Drug: tafasitamab; Drug: parsaclisib
- Part 4: tafasitamab combination therapy (Experimental): tafasitamiab in combination with lenalidomide will be further evaluated in Group 6 at RP2D determined in Part 2.
  Interventions: Drug: tafasitamab; Drug: lenalidomide

INTERVENTIONS:
Drug: tafasitamab — tafasitamab will be administered at protocol defined timepoints based on the groups participants are assigned.
  Other Names: INCMOR00208; MOR00208; Xmab5574
Drug: lenalidomide — lenalidomide will be administered orally at protocol defined timepoints based on the groups participants are assigned.
  Arms: Part 2 : tafasitamab combination therapy; Part 4: tafasitamab combination therapy
Drug: parsaclisib — parsaclisib will be administered at protocol defined timepoints based on the groups participants are assigned.
  Arms: Part 2 : tafasitamab combination therapy; Part 3 : Dose Expansion of tafasitamab +parsaclisib
Drug: R-CHOP — R-CHOP is a combination regimen consisting of rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisolone. R-CHOP will be administered at protocol defined timepoints based on the groups participants are assigned.
  Arms: Part 2 : tafasitamab combination therapy

SUMMARY:
This is an open-label, multicenter study to evaluate safety and tolerability, determine the RP2Ds of tafasitamab alone in Japanese participants with R/R NHL, or to evaluate efficacy and safety of tafasitamab in combination with lenalidomide in Japanese participants with R/R DLBCL, or tafasitimab in combination with lenalidomide plus R-CHOP in Japanese participants with previously untreated DLBC, or tafasitimab in combination with lenalidomide in Japanese participants with previously R/R DLBC.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 only: Biopsy-proven participants with relapsed or refractory NHL of DLBCL, FL or MZL.
* Groups 3, 4a and 5 only: Biopsy-proven participants with relapsed or refractory DLBCL.
* Groups 2 and 6 only: Biopsy-proven participants with DLBCL and another select lymphoid neoplasms.
* Participants must have at least 1 bi-dimensionally measurable lesion.
* ECOG performance status of 0 to 2.
* Participants with protocol defined laboratory criteria at screening as defined in the protocol.
* Group 1 only:

Received at least 1 previous systemic therapy line for the treatment of NHL. At least 1 previous therapy line must have included a CD20-targeted therapy (eg, RTX).

* Groups 2, 3, 4a and 6 only:

Received at least 1, but no more than 3, previous systemic therapy lines for the treatment of DLBCL. At least 1 previous therapy line must have included a CD20-targeted therapy (eg, RTX).

* Group 5 only: Participants must have:

  1. Untreated DLBCL.
  2. Ann Arbor Stage III to IV.
  3. IPI status of 3 to 5 or age-adjusted IPI 2-3 (in Group 5 only).
  4. Appropriate candidate for R-CHOP.
  5. LVEF of ≥ 50%, assessed by echocardiography.
* Willingness to avoid pregnancy or fathering children.
* In the opinion of investigator, the participant must:

  1. Not have a history of noncompliance in relation to medical regimens or be considered potentially unreliable and/or uncooperative.
  2. Be able to understand the reason for complying with the special conditions of the pregnancy prevention risk management plan and give written acknowledgement of this.

Exclusion Criteria:

* Any other histological type of lymphoma.
* History of prior non-hematologic malignancy.
* Congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias.
* Participants with known positive test result for hepatitis C, and hepatitis B.
* Known seropositive for or history of active viral infection with HIV.
* Known active bacterial, viral, fungal, mycobacterial, or other infection at screening.
* Known CNS lymphoma involvement - present or past medical history.
* History or evidence of clinically significant cardiovascular, CNS and/or other systemic disease that would in the investigator's opinion preclude participation in the study or compromise the participant's ability to give informed consent.
* History or evidence of rare hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.
* History or evidence of interstitial lung disease.
* Vaccination with live vaccine within 21 days prior to study treatment (Note: throughout the study treatment period and at least 6 months after end of treatment, vaccination with live vaccines should be avoided).
* Major surgery within up to 30 days prior to signing the ICF, unless the participant is recovered at the time of signing the ICF.
* Any anticancer and/or investigational therapy within 14 days prior to the start of Cycle 1.
* Groups 2, 3, 4a, 5 and 6 only: Gastrointestinal abnormalities including the inability to take oral study treatment, requiring IV alimentation, or prior surgical procedure affecting absorption.
* Pregnancy or lactation.
* Groups 2, 3, 5 and 6 only: Participants who have history of deep venous thrombosis/embolism, threatening thromboembolism, stroke or known thrombophilia or are at a high risk for a thromboembolic event in the opinion of the investigator and who are not willing/able to take venous thromboembolic event prophylaxis during the entire treatment period if required
* Group 4a only: Use or expected use during the study of any restricted medications, including potent CYP3A4 inhibitors or inducers within 14 days or 5 half-lives (whichever is longer) before the date of study treatment administration
* Groups 1, 3, 4a and 6 only: Participants who have:

  1. Not discontinued CD20-targeted therapy, chemotherapy, radiotherapy, investigational anticancer therapy, or other lymphoma-specific therapy within the 14 days prior to Day 1 dosing.
  2. In the opinion of the investigator, not recovered sufficiently from the adverse toxic effects of prior therapies.
  3. Groups 1, 3 and 4a only: Previous treatment with CD19-targeted therapy (eg, CD19-CAR-T therapies, other CD19 mAbs including bispecific and ADCs).

     Groups 2 and 6 only: Previous treatment with tafasitamab. Note: Participants in Groups 2 and 6 who have received previous CD19 directed therapy (other than tafasitamab) must have CD19-positive lymphoma confirmed by a biopsy taken after completing the prior CD19-targeted therapy.
  4. Groups 2, 3 and 6 only: Been previously treated with IMiDs (eg, thalidomide or LEN).
  5. Group 4a only: Been previously treated with selective PI3Kδ or pan-PI3K inhibitors (eg, idelalisib, copanlisib, duvelisib) and/or Bruton's tyrosine kinase inhibitors (eg, ibrutinib).
  6. A history of hypersensitivity to compounds of similar biological or chemical composition to tafasitamab, IMiDs, and/or the excipients contained in the study treatment formulations (citric acid monohydrate, polysorbate 20, sodium citrate dehydrate and trehalose dihydrate).
  7. Undergone ASCT within the period ≤ 3 months before the signing of the ICF. Participants who have a more distant history of ASCT must exhibit full hematological recovery before enrolment into the study.
  8. Undergone previous allogenic stem cell transplantation.
  9. Concurrent treatment other anticancer or experimental treatments.
* Group 5 only: Participants who have:

  1. A history of radiation therapy to ≥ 25% of the bone marrow for other diseases or history of anthracycline therapy.
  2. A history of hypersensitivity or contraindication to any component of R-CHOP, LEN, or compounds of similar biological or chemical composition as tafasitamab and/or the excipients contained in the study treatment formulations or R-CHOP.
  3. Contraindication to any of the individual components of R-CHOP.
  4. Any anticancer and/or investigational therapy within 30 days prior to the start of Cycle 1, except for permitted prephase treatment defined below.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Part 1,2 and 3 : Treatment Emergent Adverse Events (TEAE'S) | Approximately 2 years
  Adverse events reported for the first time or worsening of a pre-existing event after first dose of study treatment.
Part 4: Objective Response | Approximately 27 months
  Best Response of complete/complete metabolic response or partial/partial metabolic response

SECONDARY OUTCOMES:
Part 1,2, 3 and 4 : Cmax of tafasitamab | Approximately 27 months
  Maximum observed serum concentration.
Part 1, 2, 3 and 4: Cmin of tafasitamab | Approximately 27 months
  Minimum observed serum concentration over the dose interval.
Part 4: Complete Response | Approximately 27 months
  Defined as the proportion of participants with Complete Response as determined by an IRC and investigator assessment according to the Lugano criteria
Part 4: Duration of Response | Approximately 27 months
  Defined as the time from the date of first documented evidence of CR or PR until the first documented disease progression or death from any cause, whichever occurs first, among participants who achieve an objective response as determined by IRC and investigator assessment based on the Lugano criteria for response assessment
Part 4: Progression-Free Survival | Approximately 27 months
  Defined as the time from the date of randomization until the first documented disease progression as determined by IRC and investigator assessment based on the Lugano criteria for response assessment or death from any cause, whichever occurs first.
Part 4: Overall Survival | Approximately 27 months
  Defined as the time from the date of randomization until death from any cause.
Part 4: Overall Response Rate | Approximately 27 months
  Defined as the proportion of participants with a CR or PR as determined by the investigator based on the Lugano criteria for response assessment
Part 4: Treatment Emergent Adverse Events (TEAE'S) | Approximately 2 years
  Adverse events reported for the first time or worsening of a pre-existing event after first dose of study treatment.

CONTACTS AND LOCATIONS:
Locations (23):
- Japan (23):
  - Aichi Cancer Center Hospital, Aichi
  - Chiba Cancer Center, Chiba
  - National Cancer Center Hospital East, Chiba
  - University of Fukui Hospital, Fukui
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - Kobe City Medical Center General Hospital, Hyōgo
  - Tokai University Hospital, Kanagawa
  - The Cancer Institute Hospital of Jfcr, Kōtoku
  - Nho Kumamoto Medical Center, Kumamoto-ken
  - Nho Shikoku Cancer Center, Matsuyama
  - Tohoku University Hospital, Miyagi
  - Japanese Red Cross Nagoya Daini Hospital, Nagoya
  - Iuhw Narita Hospital, Narita
  - Nho Okayama Medical Center, Okayama
  - Saitama Medical Center, Saitama-shi
  - Nho Hokkaido Cancer Center, Sapporo
  - Kindai University Hospital, Sayama
  - Osaka University Hospital, Suita-shi
  - Nho Disaster Medical Center, Tachikawa
  - National Cancer Center Hospital, Tokyo
  - Mie University Hospital, Tsu
  - Kanagawa Cancer Center, Yokohama

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- [Derived] Izutsu K, Fukuhara N, Yuda J, Suehiro Y, Kusumoto S, Casadebaig ML, Suzukawa K, Fukushima K. Tafasitamab as Monotherapy or in Combination in Japanese Patients With B-Cell Non-Hodgkin Lymphoma: Results From the Phase 1b J-MIND Study. Cancer Sci. 2026 Jan 21. doi: 10.1111/cas.70306. Online ahead of print. PMID 41563911
- See also: To assess the safety and tolerability of tafasitamab alone or in combination with other drugs in Japanese participants with Non-Hodgkins Lymphoma (NHL) (J-MIND) — https://incyteclinicaltrials.com/studies/incmor-0208-102